CLINICAL TRIAL: NCT06202118
Title: A Pilot Feasibility and Safety Trial of Intratumoral Diffusing Alpha-emitter Radiation Therapy (DaRT) for the Treatment of Newly Diagnosed or Recurrent Breast Carcinoma in Frail or Elderly Patients.
Brief Title: A Study of Diffusing Alpha Radiation Therapy for Patients With Breast Carcinoma in Frail or Elderly Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-BRST-07
Record Dates: First submitted 2023-12-31; First posted 2024-01-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Recurrent Breast Cancer; Breast Carcinoma
Keywords: Alpha radiation; Breast cancer; Newly Diagnosed Breast Carcinoma; Breast carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of radioactive sources [Ra-224 containing stainless-steel 316LVM tubes- (Alpha DaRT seeds)]. The seeds release by recoil into the tumor short-lived alpha-emitting atoms

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for the treatment of newly diagnosed or Recurrent Breast Carcinoma in frail or elderly patients.

DETAILED DESCRIPTION:
This is a Prospective Open label Single arm multi-center interventional study. The study is designed to evaluate the Feasibility and Safety of DaRT seeds for the treatment of newly diagnosed or Recurrent Breast Carcinoma in frail or elderly patients.

The study will be comprised of a screening period, DaRT insertion visit, acute follow-up phase of 4- 8 weeks and a long-term follow up phase of 24 months. The total duration of the study will be 24 months from the DaRT insertion procedure.

A total of 10 subjects will be enrolled from all breast cancer subtypes (HR+/HER-2-, HR+/HER-2+, HR-/HER-2-, and HR-/HER-2-.). No formal interim analysis is planned for this study.

Eligible patients who meet inclusion/exclusion criteria (as assessed during the screening period) will be invited to the site for the procedure of DaRT seeds insertion. The patients will be monitored for a period of 24 months post insertion

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast tumor with no involvement of skin within 12 months.
* Tumor size ≤ 4 centimeters in the longest diameter.
* Tumor is not deemed as resectable with radical surgery or the patient does not wish to go through surgery
* De-novo or recurrent lesions.
* Single lesion per quadrant per subject.
* Targeted lesion must be technically amenable for complete coverage (including margins) by the DaRT seeds.
* Interstitial implant indication validated by multidisciplinary team.
* ECOG Performance Status ≤3.
* Life expectancy ≥12 months.
* Women Age ≥65 or younger if unfit for standard of care.
* Willing and have the ability to provide signed Informed Consent.
* Blood tests values:

  * Leucocytes ≥3000mm3,
  * Absolute neutrophil count ≥1500mm3,
  * Platelets ≥100,000 mm3,
  * Total bilirubin ≤ 1.5xULN,
  * AST, SGOT, SGPT ≤2.5xULN, If Alkaline Phosphatase ≤ 4xULN, then transaminases are normal.
  * Creatinine ≤ 2.0xULN.
  * INR or Prothrombin time ≤1.5xULN

Exclusion Criteria:

* T4 category with skin involvement.
* Ductal carcinoma in situ.
* Inflammatory breast carcinoma.
* Longest tumor diameter >4 cm.
* Patients with prior radiation to the same area within the past 6 months.
* Has a known additional malignancy that is progressing or requires active treatment.
* Patients undergoing immunosuppressive and/or systemic corticosteroid treatment except for steroid inhalations for treatment of asthma or lung disease
* Subjects not willing to sign an informed consent.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility -DaRT seed placement | immediately following the insertion procedure
  Feasibility will be determined according to the Rate of successful placement of DaRT seeds via imaging
Safety- Adverse events | From Day 0
  Safety will be determined according to the overall incidence of device related SAE'sgraded according to CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Efficacy - Control evaluation | 3,6,12 and 24 months
  To evaluate efficacy, as determined by local control evaluation according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No